CLINICAL TRIAL: NCT00532454
Title: A Clinical Study for the Evaluation of the Association Between CYP2D6 Genetic Polymorphisms and the Treatment Effect of Tamoxifen in Patients With Metastatic Breast Cancer
Brief Title: Evaluation of the Association Between CYP2D6 Genetic Polymorphisms and the Treatment Effect of Tamoxifen
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: planned to design a prospective study
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: CENTER FOR BREAST CANCER, NATIONAL CANCER CENTER
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-06-198
Record Dates: First submitted 2007-09-19; First posted 2007-09-20 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2007-09

CONDITIONS: Breast Cancer; Metastatic Disease
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tamoxifen (Other): observation for clinical efficacy on tamoxifen according to CYP2D6 genotype
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Tamoxifen — tamoxifen 20mg, PO, QD until disease progression

SUMMARY:
Primary objectives of this study is to evaluate the effects of CYP2D6 genotypes on time to progression after tamoxifen treatment in pre- or postmenopausal women with metastatic breast cancer. Furthermore, we will evaluate the effects of CYP2D6 genotypes on clinical benefit and response duration to tamoxifen administration in pre- or postmenopausal women with metastatic breast cancer and also evaluate the effects of CYP2D6 genotypes on the steady state plasma concentration of tamoxifen and its metabolites

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically diagnosed stage IV or recurrent breast cancer patients according to American Joint Committee on Cancer (AJCC)
* Positive estrogen receptor or Positive progesterone receptor.
* Females at least 18 years of age.
* Prior radiation therapy is allowed as long as the irradiated area is not the only source of measurable disease
* Prior hormone therapy less than 2.
* No history of Megace medication for recent 28 days
* Performance status of 0, 1 and 2 on the ECOG criteria
* Clinically measurable disease, defined as bidimensionally measurable lesions with clearly defined margins on x-ray, CT scan, MRI or physical examination. Lesions serving as measurable disease must be at east 1 cm by 1 cm, as defined by x-ray, CT scan, MRI, or physical examination
* Bone only or pleural fluid only disease is included as long as evaluation for clinical benefit is possible
* Estimated life expectancy of at least 12 weeks
* Compliant patient who can be followed-up adequately.
* Adequate hematologic (WBC count 3,000/mm3, platelet count 100,000/mm3), hepatic (bilirubin level 1.8 mg/dL, AST, ALT 1.5xULN, albumin 2.5 g/dL), and renal (creatinine concentration 1.5 mg/dL) function.
* Informed consent from patient or patient's relative
* Childbearing women should use non-hormonal contraceptive method

Exclusion Criteria:

* Active or uncontrolled infection.
* Second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin or prior malignancy treated more than 5 years ago without recurrence).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-06; Primary Completion 2006-06 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
efficacy of tamoxifen | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jungsil Ro, MD, PhD, Principal Investigator — National Cancer Center, Korea
Locations (2):
- South Korea (2):
  - National Cancer Center, 809 Madu1-dong, Ilsandong-gu, Goyang-si, Gyeonggi-do
  - National cancer center, Goyang-si, Gyeonggi-do